CLINICAL TRIAL: NCT02538276
Title: Study of a Real-word Registry of Carotid Endarterectomy and Carotid Artery Stenting in Brazil. Analysis of Prospective Cases of the Registry of Vascular Diseases at University Hospitals of the State of São Paulo
Brief Title: Carotid Endarterectomy and Carotid Artery Stenting in Brazil
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Edwaldo Edner Joviliano, MD; PhD, University of Sao Paulo
Other Study IDs: 01/2013
Record Dates: First submitted 2015-08-24; First posted 2015-09-02 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Arterial Diseases, Carotid
Keywords: carotid endarterectomy, carotid stenosis, carotid stenting
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group carotid endarterectomy (CEA): Patients submitted to carotid endarterectomy
- Group carotid stenting (CAS): Patients submitted to carotid artery stenting

SUMMARY:
Cerebrovascular disease is a leading cause of death and the leading cause of serious long-term disability. Carotid artery stenting (CAS) and carotid endarterectomy (CEA) are alternative strategies for stroke prevention in patients with atherosclerotic carotid disease.The safety and efficacy of CAS compared to CEA still remains questioned, and CEA has been considered to the first-line treatment of carotid stenosis in worldwide. The purpose of this study is to compare the practice and outcomes of CAS and CEA in a real world setting at Public University Hospitals in Brazil.

DETAILED DESCRIPTION:
This study will be a prospective analysis of the treatment of patients with carotid stenosis through carotid endarterectomy and carotid artery stenting performed at 5 centers proposed by five years with the Vascular Study Group from public Universities of Sao Paulo state in Brazil. The primary outcome measures will be:

1. any in-hospital stroke.
2. any stroke, death, or myocardial infarction (MI). Patients undergoing CEA in conjunction with cardiac surgery will be excluded. Multivariate logistic regression will be performed to identify predictors of stroke or death in patients undergoing CEA and CAS.

The characteristics and background of patients who underwent CAS and CEA include: age, gender, carotid endarterectomy high risk; also presentation of symptoms, and degree of stenosis will be analyzed. Next, procedural success, periprocedural antiplatelet use, embolic protection device use, the type of stent (open-cell or closed-cell) or patch to carotid, the execution of pre ballooning or post ballooning dilatation at carotid artery stenting, and procedure-related complications will be analyzed to clarify the current strategy and the treatment results of both techniques . Degree of stenosis have been measured in accordance with North American Symptomatic Carotid Endarterectomy Trial method.

Outcomes will be stratified by symptomatic and asymptomatic status. Symptomatic patients are defined as having a neurologic event, including any hemispheric or ocular transient ischemic attack,major or minor stroke preceding the intervention ipsilateral to the treated lesion. Technical success relates to periprocedural events that occur from the initiation of the procedure and extend through the first 24-hour postoperative period. Primary technical success was defined on an intent-to-treat basis, and it will requires the successful exclusion of the carotid plaque by surgical or interventional means. Technical success include the outcomes and complications of preoperative carotid angiograms whenever these imaging studies are obtained prior to the carotid intervention. For carotid endarterectomy, primary technical success implies a successful removal of the carotid plaque and closure of the artery with or without patch and less than a 30% residual stenosis. For carotid stenting, the introduction and deployment of the embolic protection device and the carotid stent in the absence of stroke, myocardial infarction, death, surgical conversion, or vascular obstruction constitutes primary technical success.

All complications should be categorized as local vascular, local nonvascular, and systemic. Other complications. As with any vascular procedures, complications after carotid interventions should be reported in a systematic and standardized manner with a description of the degrees of severity. Although assigning a degree of severity to all complications of different methods of treatment may be difficult, severity scales should be provided whenever possible so adverse events can be assessed and compared. The following severity scale has been modified from the reporting standards for lower extremity ischemia:Mild (1) refers to a complication that resolves spontaneously or with minimal intervention, does not increase the hospital length of stay, and does not cause permanent disability. Moderate (2) refers to the need for significant intervention, prolongation of hospitalization more than 24 hours, and at most, minor permanent disability that does not interfere with normal daily activity. A severe complication (3) needs major surgical, endovascular or medical intervention, may be associated with prolonged convalescence, is usually accompanied by prolonged or permanent disability, and may result in death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid stenosis > 70% who wil be underwent to carotid endarterectomy or carotid artery stenting.

Exclusion Criteria:

* Need to concomitant cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent to carotid endarterectomy (CEA)or carotida artery stenting(CAS) for treat carotid stenosis at the any of the five hospitals involved in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
any stroke | 30-day
  major or minor, ipsilateral or contralateral. Postoperative major strokes will be defined as cortical, vertebrobasilar, or ocular disability resulting in nonindependent living status, or blindness; otherwise strokes will be defined as minor

SECONDARY OUTCOMES:
any stroke, death or myocardial infarction | 30-day
  major or minor, ipsilateral or contralateral for stroke, 30-day mortality and/or myocardial infarction confirmed by electrocardiogram and / or positive marker (Troponin).

CONTACTS AND LOCATIONS:
Overall Officials: EDWALDO E JOVILIANO, MD; PHD, Principal Investigator — University of Sao Paulo
Locations (5):
- Brazil (5):
  - University Hospital of Botucatu Medical School, Botucatu, São Paulo
  - University Hospital of School of Medical Sciences UNICAMP, Campinas, São Paulo
  - University Hospital of Marilia Medical School, Marília, São Paulo
  - University Hospital of Ribeirao Preto Medical School, University of São Paulo, Ribeirão Preto, São Paulo
  - University Hospital of São Jose do Rio Preto Medical School, São José do Rio Preto, São Paulo

REFERENCES:
- [Derived] Joviliano EE, Ribeiro MS, Sobreira ML, Moura R, Geiger MA, Guillamon AT, Regina de Oliveira Raymundo S, Miquelin DG, Hafner L, Almeida MJ, Oliveira TF, Dalio MB, Yoshida WB. Short-Term Outcomes of Transfemoral Carotid Artery Stenting and Carotid Endarterectomy in Symptomatic Patients: Data from a Multicentric Prospective Registry in Brazil. Ann Vasc Surg. 2022 Sep;85:41-48. doi: 10.1016/j.avsg.2022.04.053. Epub 2022 May 16. PMID 35589029
- [Derived] Joviliano EE, Yoshida WB, Sobreira ML, Moura R, Guillaumon AT, Raymundo SR, Miquelin DG, Hafner L, Almeida MJ. An Observational Registry of Carotid Endarterectomy and Carotid Artery Stenting in Brazil: Study Protocol. JMIR Res Protoc. 2016 Nov 23;5(4):e226. doi: 10.2196/resprot.5986. PMID 27881360